CLINICAL TRIAL: NCT06333821
Title: A Multicentre, Prospective, Randomized, Double-blind, Placebo-controlled Study of Nimotuzumab Plus Concurrent Chemoradiotherapy Sequential Maintenance Treatment for Locally Advanced Cervical Squamous Cell Carcinoma
Brief Title: A Study of Nimotuzumab Plus Concurrent Chemoradiotherapy Sequential Maintenance Treatment for Cervical Carcinoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biotech Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BPL-Nim-CC-3003
Record Dates: First submitted 2023-02-09; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — nimotuzumab; Cisplatin; Brachytherapy

STUDY DESIGN:
Intervention Model Description: This is a multicenter prospective, randomized, double-blind, placebo-controlled phase III trial
Who Masked: Participant, Investigator
Masking Description: This study is double-blind and will blind both the investigator and the subjects. All participants in the study (including data managers and biostatisticians) will be unaware of treatment assignment (except blind statisticians).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nimotuzumab+chemoradiotherapy (Experimental): Participants receive Nimotuzumab 400 mg intravenously (IV) on Day 1 of each week cycle (QW) for 7-8 cycles followed by Nimotuzumab 400 mg IV on Day 1 of each 2-week cycle (Q2W) for an additional 12 cycles. During the QW dosing period of Nimotuzumab, participants receive concurrent chemoradiotherapy. The standard of care chemoradiotherapy regimen includes cisplatin 40 mg/m^2 IV once or divides into 3 times per week (QW) for 4 or 5 weeks plus external beam radiotherapy (EBRT) followed by brachytherapy with minimum total radiotherapy dose of 80-85 Gray Units (Gy) for volume-directed given with the total duration of radiation treatment not to exceed 8 weeks .
  Interventions: Biological: Nimotuzumab; Drug: Cisplatin; Radiation: External Beam Radiotherapy (EBRT); Radiation: Brachytherapy
- placebo for Nimotuzumab+chemoradiotherapy (Experimental): Participants receive placebo for Nimotuzumab 400 mg intravenously (IV) on Day 1 of each week cycle (QW) for 7-8 cycles followed by placebo 400 mg IV on Day 1 of each 2-week cycle (Q2W) for an additional 12 cycles. During the QW dosing period of placebo, participants receive concurrent chemoradiotherapy. The standard of care chemoradiotherapy regimen includes cisplatin 40 mg/m^2 IV once or divides into 3 times per week (QW) for 4 or 5 weeks plus external beam radiotherapy (EBRT) followed by brachytherapy with minimum total radiotherapy dose of 80-85 Gray Units (Gy) for volume-directed given with the total duration of radiation treatment not to exceed 8 weeks .
  Interventions: Drug: Cisplatin; Radiation: External Beam Radiotherapy (EBRT); Radiation: Brachytherapy; Drug: placebo for Nimotuzumab

INTERVENTIONS:
Biological: Nimotuzumab — Nimotuzumab 400mg
  Arms: Nimotuzumab+chemoradiotherapy
Drug: Cisplatin — Cisplatin 40mg/m^2
Radiation: External Beam Radiotherapy (EBRT) — External Beam Radiotherapy (EBRT)
Radiation: Brachytherapy — Brachytherapy
Drug: placebo for Nimotuzumab — placebo for Nimotuzumab 400mg
  Other Names: placebo
  Arms: placebo for Nimotuzumab+chemoradiotherapy

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of nimotuzumab plus concurrent chemoradiotherapy sequential maintenance therapy versus placebo combined with concurrent chemoradiotherapy in patients with locally advanced cervical squamous cell carcinoma.

The primary hypotheses are that nimotuzumab plus concurrent chemoradiotherapy sequential maintenance therapy is superior to placebo plus concurrent chemoradiotherapy with respect to progression-free survival.

DETAILED DESCRIPTION:
This is a multicenter, prospective, randomized, double-blind, placebo-controlled clinical study.The trail will enroll 460 subjects (FIGO 2018, stageIB3-IVA)who meet enrollment criteria but do not meet exclusion criteria. According to clinical stage (FIGO 2018 stage, stage IB3-IIB or III-IVA) 、tumor diameter (>4cm or ≤4cm)、 age (≥18 years and < 65 years old or ≥65 years old and ≤80 years old) for stratified randomization. They are divided into experimental group and control group according to 1:1. Patients in the experimental group will receive nimotuzumab 400mg on the basis of concurrent chemoradiotherapy, once a week for 7-8 weeks, and then maintenance treatment once every 2 weeks for 24 weeks. Using placebo(Nimotuzumab injection mimics) in the control group 80 ml on the basis of concurrent chemoradiotherapy, once a week for 7 to 8 weeks, after the maintenance treatment, once every 2 weeks for 24 weeks. Patients with incomplete tumor response assessed by imaging and pathological examination 3 months after radiotherapy can be given 2-4 cycles of adjuvant chemotherapy with cisplatin/carboplatin combined with paclitaxel regimen. Regular imaging examination and survival follow-up were performed after treatment. The primary efficacy end point was progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

* 1.Aged 18-80 years old;
* 2.Histologically diagnosed primary cervical squamous cell carcinoma, with clinical stage IB3-IVA (FIGO 2018);
* 3.At least one measurable lesion according to RECIST 1.1;
* 4.Absence of severe hematopoietic dysfunction and heart, lung, liver, kidney dysfunction and immunodeficiency, laboratory test results meet the following criteria: Hemoglobin ≥ 90 g/L; Absolute neutrophil count ≥ 1.5 × 10^9/L and white blood cell count ≥ 3.0 × 10^9/L; Platelet count ≥ 100 × 10^9/L; Aspartate aminotransferase (AST) ≤ 2.5 × ULN; Alanine aminotransferase (ALT) ≤ 2.5 × ULN ; Total bilirubin ≤ 1.5 × ULN; Serum creatinine ≤ 1.0 × ULN;
* 5.ECOG score 0-1 points;
* 6.Women of childbearing potential must have a negative serum or urine HCG within 72 hours prior to enrollment (postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential. A pregnancy test is not required for women who have demonstrated tubal ligation); Women of childbearing potential who are willing to take medically recognized contraceptive measures during the trial;
* 7.Compliance is good and informed consent is voluntarily signed.

Exclusion Criteria:

* 1.Cervical adenocarcinoma and rare pathological types of malignant tumors;
* 2.Previous surgery for cervical cancer, pelvic radiation therapy, systemic chemotherapy, tumor targeted therapy, immunotherapy;
* 3.Ureteral obstruction, inability to place ureteral stent or pyelostomy;
* 4.Pregnant or lactating women;
* 5.Patients with rectovaginal fistula/vaginovesical fistula/uncontrolled vaginal bleeding or at risk of fistula;
* 6.Had undergone major surgery (except biopsy) within 4 weeks prior to randomization;
* 7.Had received a live vaccine within 4 weeks prior to the initial study drug treatment or planned to vaccinate during the study;
* 8.Human immunodeficiency virus (HIV) infection;Active hepatitis B (the quantitative detection result of HBV DNA exceeds the lower limit of detection), or HCV infection (the quantitative detection result of HCV RNA exceeds the lower limit of detection);
* 9.Had the following serious medical conditions: a) Uncontrolled hypertension (defined as systolic blood pressure > 150 mmHg or diastolic blood pressure > 100 mmHg), or had experienced a hypertensive crisis; b) Myocardial infarction and unstable angina occurred within 6 months before randomization; c) Decompensated heart failure within three months before enrollment (NYHA class III and IV); d) The presence of severe arrhythmias requiring long-term medical intervention, except in patients with asymptomatic atrial fibrillation with stable ventricular rate; e) Left ventricular ejection fraction (LVEF)<50%; f) The presence of uncontrolled hyperglycemia; g) The presence of uncontrollable infections；
* 10.The presence of active or suspected autoimmune diseases, except for type 1 diabetes、hypothyroidism or skin conditions that do not require systemic treatment (vitiligo、psoriasis or alopecia)；
* 11.Conditions requiring systemic treatment with corticosteroids or other immunosuppressive agents within 14 days before randomization；
* 12.Patients with a history of other malignant tumors (except cured cutaneous basal cell carcinoma);
* 13.Patients with Crohn's disease and ulcerative colitis;
* 14.Patients who are participating in other clinical trials or have stopped clinical trials for less than 4 weeks;
* 15.Patients with known hypersensitivity to Nimotuzumab or its components;
* 16.Patients with contraindications to cisplatin、carboplatin and paclitaxel;
* 17.Patients with neurological or psychiatric disorders affecting cognitive ability;
* 18.Patients whose lesions cannot be treated with intracavitary radiotherapy as assessed by the investigator;
* 19.Any condition that, in the opinion of the Investigator, may be inappropriate for patients in the study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2030-04-01 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed Blinded Independent Central Review (BICR) | Up to approximately 5 years
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by by the Investigator | Up to approximately 5 years
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first.
3-,5-Year Overall Survival (OS) | Up to approximately 3 and 5 years
  OS is the time from randomization to death due to any cause.
3-,5-Year Disease Free Survival(DFS) | Up to approximately 3 and 5 years
  DFS is defined as the time from randomization to disease recurrence or death due to any cause.
3-,5-Year Locoregional Recurrence-Free Survival(LRRFS) | Up to approximately 3 and 5 years
  Locoregional recurrence-free survival (LRRFS) was defined as the absence of either consistent or relapsed disease at the primary tumor site or the regional lymph nodes
3-,5-Year Distant Metastasis-free Survival (DMFS) | Up to approximately 3 and 5 years
  Distant metastasis-free survival (DMFS) was calculated from the date of patient recruitment to the date of distant metastasis.
Tumor Regression Rate(TRR) | From date of randomization until the date of brachytherapy,assessed up to 5 weeks
  The maximum diameter represents the size of the tumor by MRI. Tumor size for each patient were obtained: pre-RT tumor size (V1), pre- brachytherapy tumor size (V2). TRR=(V1-V2)/V1 × 100%.
Complete Response Rate | From date of randomization until the date of brachytherapy,assessed up to 5 weeks
  The proportion of subjects with the best complete response in this group assessed by MRI.
Complete Response Rate | 3 months later after treatment
  The proportion of subjects with the best complete response in this group assessed by MRI.
Objective Response Rate | 3 months later after treatment
  The proportion of subjects with the best complete response or partial response in this group assessed by MRI.
Change from Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Global Health Status Score | Baseline and up to approximately 5 years
  The EORTC QLQ-C30 is a questionnaire that rates the overall quality of life in cancer participants. The first 28 questions use a 4-point scale (1=not at all to 4=very much) for evaluating function (physical, role, social, cognitive, emotional), symptoms (diarrhea, fatigue, dyspnea, appetite loss, insomnia, nausea/vomiting, constipation, and pain) and financial difficulties. The last 2 questions use a 7-point scale (1=very poor to 7=excellent) to evaluate overall health and quality of life. Global scores are converted to a score of 0 to 100, with a higher score indicating improved health status. The change from baseline in EORTC QLQ-C30 score will be presented.
Change from Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Symptom Specific Scale for Cervical Cancer (EORTC QLQ-CX24) Score | Baseline and up to approximately 5 years
  The EORTC QLQ-CX24 is a questionnaire that rates the symptoms common to women with cervical cancer and evaluates the impact of disease and/or treatments. The 24 items use a 4-point scale (1=not at all to 4=very much) and are classified into 3 multi-item scales, 11 items with symptom experience, 3 items with body image, and 4 items with sexual/ vaginal functioning. The other items of the questionnaire are lymphedema, peripheral neuropathy, menopausal symptom, sexual worry, sexual activity, and sexual enjoyment. The change from baseline in EORTC QLQ-CX24 score will be presented.
Incidence of Treatment-Emergent Adverse Events | Within 30 days from the start of treatment to the end of the last treatment
  Safety was assessed as adverse events during treatment, the incidence of various adverse events such as adverse events related to the study drug during treatment, laboratory tests, etc

CONTACTS AND LOCATIONS:
Overall Officials: Junjie Wang, Study Chair — Peking University Third Hospital; Lichun Wei, Study Chair — TThe First Affiliated Hospital，the Air Force Medical University; Lijuan Zou, Study Chair — The Second Affiliated Hospital of Dalian Medical University; Zi Liu, Study Chair — First Affiliated Hospital Xi'an Jiaotong University; Jiayi Chen, Study Chair — Ruijin Hospital; Huijun Cheng, Study Chair — Henan Cancer Hospital; Rutie Yin, Study Chair — West China Second University Hospital; Xiangkun Yuan, Study Chair — Cangzhou Hospital of Integrated Traditional Chinese and Western Medicine.HeBei; Hui Qiu, Study Chair — Zhongnan Hospital; Hong Zhu, Study Chair — Xiangya Hospital of Central South University; Tiejun Wang, Study Chair — Second Hospital of Jilin University; Xiaomei Fan, Study Chair — The Fourth Hospital of Hebei Medical University Hebei Tumor Hospital; Keqiang Zhang, Study Chair — Hunan Cancer Hospital; Dihong Tang, Study Chair — Hunan Cancer Hospital; Qiongyu Lan, Study Chair — Second Affiliated Hospital of Nanchang University; Xiaoying Xue, Study Chair — The Second Hospital of Hebei Medical University; Song Gao, Study Chair — Shengjing Hospital; Guang Li, Study Chair — First Hospital of China Medical University; Qiuhong Tian, Study Chair — The First Affiliated Hospital of Nanchang University; Guoqing Wang, Study Chair — Shanxi Provincial Cancer Hospital; Dong Qian, Study Chair — The First Affiliated Hospital of USTC (Anhui Provincial Hospital); Manbo Cai, Study Chair — The First Affiliated Hospital of University of South China; Yuhua Gao, Study Chair — Liaoning Cancer Hospital & Institute; Dehua Wu, Study Chair — Nanfang Hospital, Southern Medical University; Xiaoge Sun, Study Chair — The Affiliated Hospital of Inner Mongolia Medical University; Yunyan Zhang, Study Chair — Cancer Hospital Affiliated to Harbin Medical University; Kun Gao, Study Chair — Guangxi Medical University Cancer Center; Qin Lin, Study Chair — The First Affiliated Hospital of Xiamen University; Qin Xu, Study Chair — Fujian Cancer Hospital; Hao Yang, Study Chair — Peking University Cancer Hospital Inner Mongolia Hospital; Rong Huang, Study Chair — First People's Hospital of Foshan; Xianming Li, Study Chair — Shenzhen People's Hospital; Juntao Ran, Study Chair — LanZhou University; Xiaojie Ma, Study Chair — Afﬁliated Hospital of North Sichuan Medical College; Xingrao Wu, Study Chair — Yunnan Cancer Hospital; Yipeng Song, Study Chair — Yantai Yuhuangding Hospital; Jun Wang, Study Chair — Tianjin Cancer Hospital Airport Hospital; Dapeng Li, Study Chair — Shandong Cancer Hospital ＆ Institute; Siyuan Zeng, Study Chair — Jiangxi Maternal and Child Health Hospital; Hongyun Shi, Study Chair — Affiliated Hospital of Hebei University; Weihu Wang, Study Chair — Peking University Cancer Hospital & Institute; Jidong Zhang, Study Chair — Shanxi Province Cancer Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wei S, Li X, Liu Z, Wei L, Zou L, Zhang Y, Sun X, Gao Y, Zhuo Y, Zhang M, Qu A, Zhang H, Guo H, Jiang P, Wang J. Nimotuzumab plus concurrent chemoradiotherapy sequential maintenance treatment for locally advanced cervical squamous cell carcinoma (NOTABLE-306): a multicenter, prospective, randomized, double-blind, placebo-controlled trial. J Gynecol Oncol. 2025 Dec 11. doi: 10.3802/jgo.2026.37.e46. Online ahead of print. PMID 41514314